CLINICAL TRIAL: NCT04314492
Title: Intracapsular Tonsillectomy in the Treatment of Obstructive Sleep Apnea in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Jaakko Piitulainen, Consultant, Doctor of Medical Science, Turku University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T62/2020
Record Dates: First submitted 2020-03-13; First posted 2020-03-19 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Tonsillar Hypertrophy; Sleep Apnea, Obstructive
Keywords: tonsil surgery; tonsillectomy; obstructive sleep apnea; coblation; intracapsular
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Tonsillectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intracapsular tonsillectomy with coblation (Experimental): (Total) Intracapsular tonsillectomy (ICTE) with coblation
  Interventions: Procedure: Tonsillectomy

INTERVENTIONS:
Procedure: Tonsillectomy — Intracapsular removal of tonsillar tissue (>90%) with coblation

SUMMARY:
Treating sleep apnea in adults caused by tonsillar hypertrophy with intracapsular tonsillectomy by coblation

DETAILED DESCRIPTION:
The investigators aim to study if good surgical results can be achieved by intracapsular tonsillectomy with coblation while monitoring safety, efficiency and cost-effectiveness. In adult tonsil surgery, the current practice in Finland is commonly extracapsular tonsillectomy with monopolar electrosurgery.

ELIGIBILITY:
Inclusion Criteria:

* age 16-64
* Planned tonsil surgery with informed concent
* Obstructive sleep apnea (AHI > 15)
* Tonsillar size of 3-4 on the Friedman scale

Exclusion Criteria:

* BMI > 35 (Based on finnish Käypä Hoito -recommendations)
* Central sleep apnea
* Weight loss of more than 10% within the study period
* Untreated obstruction of nasal breathing
* Treated peritonsillar abscess <1 month before enrollment
* Active tonsillar infection
* Previous tonsillar surgery (excluding incision of abscess)
* Malignancy
* High use of analgesics >1 DDD daily during last 4 weeks
* Untreated reflux
* Anticoagulative medication
* Any condition of hemophilia
* Pregnancy, lactation
* Other, evaluated by treating physician

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Apnea-hypopnea index | 6 months
  Post-operative apnea-hypopnea index reduction by 50% compared to preoperative values in polysomnography.

SECONDARY OUTCOMES:
Quality of life measured by Glasgow Benefit Inventory | 6 months and 24 month and 60 months
  General quality of life questionnaire. 18 questions, score 1-5 in each question, higher is better.
Quality of life measured by Nordic tonsil surgery register questionnaire | 6 months - up to 5 years
  Questions regarding postoperative complications and perceived symptom relief after 180 days. Yes/no questions and open questions, no score.
Quality of life measured by Epworth sleepiness scale | 6 months - up to 5 years
  Questions regarding sleepiness. Score 0-24, lower is better.
Post-operative recovery | 21 days
  Recovery speed defined as score 3 or less at rest; or 5 or less without regular analgesics use, questionnaire used: Brief Pain Inventory.
Total recovery of obstructive sleep apnea | 6 months and 24 months and 60 months
  Defined by apnea-hypopnea index <5 post-operatively in polysomnography.
Regrowth of tonsillar tissue | Pre-operative to 6 months
  Measured by photography, Friedman scale (0-4, lower is smaller).
Apnea-index | 6 months and 24 months and 60 months
  Post-operative apnea index reduction by 50% compared to preoperative values in polysomnography.
Snoring time | 6 months and 24 months and 60 months
  Post-operative reduction of snoring time in preoperative polysomnography compared to post-operative values in

OTHER OUTCOMES:
Apnea-hypopnea index | 24 months
  Post-operative apnea-hypopnea index reduction by 50% compared to preoperative values in polysomnography.
Apnea-hypopnea index | 60 months
  Post-operative apnea-hypopnea index reduction by 50% compared to preoperative values in polysomnography.

CONTACTS AND LOCATIONS:
Overall Officials: Jussi Jero, Professor, Study Director — University of Turku; Jaakko Piitulainen, M.D., Ph.D., Principal Investigator — Turku University Hospital
Locations (2):
- Finland (2):
  - Satasairaala, Pori, Satakunta
  - Turku University Hospital, Turku, Southwest Finland

IPD SHARING:
Plan to Share IPD: No